CLINICAL TRIAL: NCT04709419
Title: Study to Evaluate Celliant Diabetic Medical Socks to Increase Tissue Oxygenation and Incidence of Complete Wound Closure in Diabetic Foot Wounds
Brief Title: Celliant Socks to Increase Tissue Oxygenation and Complete Wound Closure in Diabetic Foot Wounds
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to enroll
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Hologenix, LLC (Industry)
Responsible Party: Principal Investigator, Larry Lavery, Professor and Director of Research, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU-2020-1386
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Active and Control samples will be prepared in sealed and labeled as A or B Randomization envelopes (A&B) will be provided to the research staff and used to obtain randomization assignment. After run-in evaluation subjects who continue to meet all inclusion and no exclusion criteria will be randomized in a 1:1 ratio to be treated with either Control or Celliant therapies, stratified by wound size (greater than size of 4 cm2) and study center. Study staff will use the randomization number labels and sock assignment of socks A or B contained in the envelope. The number will become the subject ID. The research staff will note the randomization number and the treatment assignment letter (A or B) on the CRF. The key, indicating therapy assignments (Active or Control), will only be available to staff not directly involved in the study until after the subject has completed study activities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Celliant Sock (Experimental): Celliant® Diabetic Medical Socks ("Celliant Socks") are intended to provide infrared radiation (IR) to increase tissue oxygen thereby increasing blood flow and circulation in the affected area leading to an effect on wound closure outcomes and possible pain reduction. Celliant® fibers are comprised of a proprietary blend of infrared (IR) emitting ceramic materials mixed with polyethylene terephthalate (PET). The proprietary blend consists of the following components: alumina oxide; silicon dioxide; and titanium dioxide. The Celliant fibers are woven or knitted into yarn and used to manufacture the Celliant Sock. The Celliant Sock content will be 82% Celliant polyester, 13% Nylon and 5% Spandex. Celliant fibers absorb energy (heat) generated by the wearer's body by radiation, convection and conduction, and also from the environment, and re emit the energy as infrared radiation back into the wearer's body.
  Interventions: Device: Celliant Diabetic Medical Socks
- Control Sock (Sham Comparator): The Control Sock will be visually identical to the Active Celliant® Sock. The sock will be made of identical materials without the Celliant® components. The Control sock will be 82% standard polyester, 13% Nylon, and 5% Spandex.
  Interventions: Device: Control (placebo) Medical Socks

INTERVENTIONS:
Device: Celliant Diabetic Medical Socks — Celliant® Diabetic Medical Socks ("Celliant Socks") are intended to provide infrared radiation (IR) to increase tissue oxygen thereby increasing blood flow and circulation in the affected area leading to an effect on wound closure outcomes and possible pain reduction.
  Arms: Celliant Sock
Device: Control (placebo) Medical Socks — The Control Sock will be visually identical to the Active Celliant® Sock. The sock will be made of identical materials without the Celliant® components. The Control sock will be 82% standard polyester, 13% Nylon, and 5% Spandex.
  Arms: Control Sock

SUMMARY:
This study is a prospective, multicenter, double-blind, 1:1 randomized clinical trial. The purpose of this study is to demonstrate that the use of Celliant Socks increases tissue oxygenation (via oxygen saturation, StO2) and incidence of wound closure in subjects with diabetic foot ulcers. This study will use hyperspectral imaging and wound assessment to measure these outcomes. The study will enroll 254 evaluable subjects total, 127 per arm to meet the Primary Endpoint. Enrollment may continue up to twenty-five hundred (2500) evaluable subjects total to meet the Key Secondary Endpoint of complete wound closure.

DETAILED DESCRIPTION:
Screening and Enrollment

Patients who present to the investigator's institution (through clinic admission, direct transfer from another facility, or through the emergency room) may be recruited to participate in the study. No direct marketing for subject recruitment will be done.

Patients approached for study participation will be at least 22 years of age at the time of consent, will undergo wound assessment, and meet all eligibility requirements. Those meeting eligibility criteria for the study will have the study explained to them by the Investigator. An Informed Consent Form will be provided to sign according to Section 11 prior to undergoing any study procedures. Patients will be encouraged to ask questions of the investigators. It will be made clear to the patient that not participating in the study will in no way influence the treatment plan or the relationship with the physician.

Wound Selection

Only one wound per subject will be included in the study. Subjects with multiple wounds will have each wound measured for volume. The wound with the largest volume meeting all eligibility requirements will be chosen for inclusion in the study. The etiology of the chosen wound, and if it is a new or recurring, will be documented.

Randomization and Blinding Procedure

Prior to study initiation, Active and Control samples will be prepared in sealed and labeled as A or B, also randomization envelopes will be provided to the research staff and used to obtain randomization assignment. Within each randomization envelope, there is an assignment of A or B. After run-in evaluation, the subjects wound will be debrided and dressed with SOC. At the end of the procedure, subjects who continue to meet all inclusion and no exclusion criteria will be randomized in a 1:1 ratio to be treated with either Control or Celliant therapies, stratified by wound size (greater than size of 4 cm2) and study center. Study staff will use the randomization number labels and sock assignment of socks A or B contained in the envelope. The number will become the subject ID. The research staff will note the randomization number and the treatment assignment letter (A or B) on the CRF. The key, indicating therapy assignments (Active or Control), will only be available to staff not directly involved in the study until after the subject has completed study activities.

Visit Schedule

Study procedures for each phase of study are outlined below. In a later section, details on each study procedure are described, including equipment designation.

Screening

1. Explain purpose and nature of the study and obtain signature on the informed consent document.
2. Screen the subject against protocol inclusion and exclusion criteria, including all pertinent tests

   1. ABI and/toe pressure
   2. Ulcer History, measurement, and classification
   3. Urine Pregnancy test (if indicated)

Baseline (may be done as same day as screening procedures)

1. Obtain general medical history and demographic information and social history
2. Complete a physical examination, body weight, height, and vital signs, including measurement of resting heart rate, respiratory rate, and blood pressure while seated.
3. Select the target ulcer
4. Obtain complete history pertinent to DFU disease including duration of the target ulcer, previous and current treatment.
5. Perform debridement if indicated. Debridement is to be performed using curette, scissors, scalpel, or forceps.
6. Perform standardized photography and measurement of the study wound (eKare or available camera with ruler). Assess the post-debridement ulcer area (cm2), perimeter (cm), and greatest depth (cm) using the inSight device (eKare, Fairfax, VA). These values are the baseline measurements for assessing accelerated wound closure at the two-week run-in visit.
7. Perform baseline SPP (note - this procedure does not need to be performed at baseline visit and can be performed at any visit through Run-In week 2/Therapy initiation visit).
8. Perform baseline tcpO2 (note - this procedure does not need to be performed at baseline visit and can be performed at any visit through Run-In week 2/Therapy initiation visit).
9. Perform baseline hyperspectral imaging assessment on the dorsal and plantar aspects of the foot.
10. Perform neuropathy and pain assessment.
11. Obtain blood for hematology, blood chemistry, etc that were not covered in inclusion/exclusion studies.
12. Subjects who do not meet eligibility and fail to qualify to enter the Run-in will be deemed Screen failures and discharged, noting the reasons for disqualification.
13. Collect all relevant concomitant medication (antibiotics, antifungals and other anti-infective therapies)
14. Wounds will be dressed SOC and offloaded per physician discretion.
15. Subjects who qualify to enter the run-in will be instructed to refrain from using excluded medications and return to the office for Run-in Visit 2 within 7 (±1) days.

Run-In Procedures/Therapy Initiation

Week 1 Run-in:

1. Assess target ulcer.
2. Perform debridement if indicated. Debridement is to be performed using a curette, scissors, scalpel, or forceps.
3. Perform standardized photography of the study wound.
4. Assess the post-debridement ulcer area (cm2), perimeter (cm), and greatest depth (cm) using the inSight device.
5. If wound size (ulcer area) increases/decreases by 30% or more, patient will be deemed a screen failure and removed from the study.
6. If wound size (ulcer area) decreases by less than 30%, patient wound will be treated with standard of care and return for run-in Week 2 Run-In within 7 (±1) days.
7. Perform hyperspectral imaging assessment on the dorsal and plantar aspects of the foot.
8. Perform pain assessment.
9. Collect all relevant concomitant medication (antibiotics, antifungals and other anti-infective therapies)
10. Wounds will be dressed SOC and offloaded per physician discretion.

Week 2 Run-in/Therapy Initiation:

1. Assess target ulcer
2. Perform debridement if indicated. Debridement is to be performed using curette, scissors, scalpel, or forceps.
3. Perform standardized photography of the study wound.
4. Assess the post-debridement ulcer area (cm2), perimeter (cm), and greatest depth (cm) using the inSight device.
5. If wound size (ulcer area) increases/decreases by 30% or more, patient will be deemed a screen failure and removed from the study.
6. If wound size (ulcer area) increases/decreases by less than 30%, patient wound will enter the study and randomized to either the Celliant Active or Control treatment arm.
7. Perform hyperspectral imaging of the dorsal and plantar aspects of the foot
8. Perform pain assessment.
9. Collect all relevant concomitant medication
10. Wound will be dressed with SOC and either Celliant Active or Control Sock applied.
11. Wound will be offloaded.
12. Provide subject with any additional medical socks needed until the next visit. Instruct the subject to change the socks if they become wet, soiled, or bloody and under any conditions dictated by PI instructions.

Therapy/Treatment Phase

Study Visit 1-11:

1. Document study compliance information from the subject

   1. Amount of time the sock was worn throughout the week
   2. Was it worn during the day/night?
   3. When/why the sock was changed.
   4. Has the sock been on in the 3 hours leading up to the appointment?
2. Remove sock and dressing and immediately perform hyperspectral imaging of the dorsal and plantar aspects of the foot if wound is active or closed.
3. Assess target ulcer (if wound has closed, document as such, perform steps 7 and 8 and skip to Study Visit - Wound Closed).
4. Debridement is to be performed, if indicated, using curette, scissors, scalpel, or forceps. If debridement is necessary at weekly visits, all therapy must be removed and replaced post-debridement.
5. Perform standardized photography of the study wound.
6. Assess the ulcer area (cm2), perimeter (cm), and greatest depth (cm) using the inSight device - if the wound is deemed closed by the physician, skip to EOS visit.
7. Perform SPP and tcPO2 measurements at Visit 4 (maybe be taken instead at visit 5 or 6 if subject has not been wearing their treatment sock leading up to the visit or misses this visit).
8. Collect all relevant concomitant medication
9. Perform pain assessment.
10. Redress the wound with standard of care (if wound is still active) and apply Celliant Active or Control Sock and apply offloading (if indicated).
11. Wound will be offloaded.
12. Provide subject with any additional medical socks needed until the next visit. Instruct the subject to change the socks if they become wet, soiled, or bloody and under any conditions dictated by PI instructions. Instruct the subject that they must wear the sock at all times and that including the 3 hours leading up to the next study visit.

Study Visit - Wound Closed

1. The study wound is defined as closed when there is complete skin re-epithelialization without drainage or dressing requirements confirmed by the evaluating physician at 2 consecutive study visits 2 weeks apart.
2. At this visit the subject will perform the EOS evaluation and enter the follow-up phase of the study.

Study Visit 12/EOS

1. If the study wound closes prior to the 12-week study mark, subjects will perform EOS visit at the time of wound closure. See Study Visit - Wound Closed.
2. A subject whose wound does not close completely by week 12 will exited from the study after the week 12 wound evaluation.
3. Document study compliance information from the subject

   1. Amount of time the sock was worn throughout the week
   2. Was it worn during the day/night?
   3. When/why the sock was changed.
   4. Has the sock been on in the 3 hours leading up to the appointment?
4. Remove sock and dressing and immediately perform hyperspectral imaging of the dorsal and plantar aspects of the foot if wound is active or closed.
5. Assess target ulcer (if wound has closed, document as such, perform steps 7-12 and skip to Study Visit - Wound Closed).
6. Perform standardized photography of the study wound.
7. Assess the ulcer area (cm2), perimeter (cm), and greatest depth (cm) using the inSight device.
8. Perform SPP if wound is active or closed.
9. Perform tcpO2 if wound is active or closed.
10. Perform pain assessment
11. Ask the subject if they thought they were in the active or control group
12. Administer DFS-SF
13. Collect all relevant concomitant medication
14. Redress the wound per physician-directed standard of care.

Study Visit Follow up

1. If the subject's wound closes within the 12-week treatment window, they will enter the follow up phase of the study.
2. At 3 months post closure, wound evaluation will be performed as outlined below. This followup visit will be in person. In the event that an in-person visit is not possible, a telehealth visit may be performed and documented as such.:

   a. Assess the study wound to determine that it remained closed b. If the study wound has reoccurred i. record the date of reoccurrence ii. measure the size of dehiscence or re-ulceration iii. exit the subject from the follow up phase c. Assess the study foot for new sites of ulceration i. record the date of reoccurrence ii. measure the size of dehiscence or re-ulceration iii. exit the subject from the follow up phase

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus
* Subject is willing and able to wear a sports-style tube sock at least 22 hours a day.
* Ankle Brachial Index (ABI) ≥0.5 (bedside ABI is acceptable for screening purposes as the formal imaging ABI may not be resulted prior to surgery) or toe pressure of ≥30mmHg
* One or more diabetic foot ulcers (only one will be treated) that are located in the ankle area or below that has persisted a minimum of 30 days prior to the Screening visit
* Diabetic Foot Ulcers ≥1cm2 and ≤16cm2
* Ulcer grade I or II, Stage A, I or II Stage B, according to University of Texas Wound Classification System
* 22 years of age or older

Exclusion Criteria:

* Has clinically significant renal disease to require hemo or peritoneal dialysis
* Subject has untreated osteomyelitis
* Ulcers within 5cm of target ulcer or connected by fistulas
* Ulcer has decreased by 30% or more at the end of the run-in period
* Subject has untreated cellulitis
* Subject has untreated charcot
* Major immunodeficiency including HIV
* Is pregnant or plans to become pregnant
* Is nursing or actively lactating
* Developmental disability/significant psychological disorder that in the opinion of the investigator could impair the subject's ability to provide informed consent, participate in the study protocol or record study measures, including untreated schizophrenia, bipolar disorder and psychiatric hospitalization within the last 2 years.
* Active alcohol or substance abuse in the opinion of the investigator that could impair the subject's ability to provide informed consent, participate in the study protocol or record study materials

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A Lavery, DPM MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total protocol enrollment was 4 subjects. 3 of which were screen fails and 1 was withdrawn by the PI.
Pre-assignment Details: 3 subjects screen failed before assignment to groups. 1 subject was assigned to the experimental arm.
Period: Overall Study
Arm/Group | Celliant Sock | Control Sock
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Total protocol enrollment was 4 subjects. 3 of which were screen fails and 1 that was assigned on the experimental arm did not complete the study and was withdrawn by the PI.
Groups:
- Total: Total of all reporting groups
Arm/Group | Celliant Sock | Control Sock | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian- Non Hispanic | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Tissue Oxygenation
Description: To compare the percent change from baseline in tissue oxygenation in Celliant and Control treated groups as measured by hyperspectral imaging.
Time Frame: 12 weeks
Population: The study duration of the only enrolled participant and withdrawn was only 79 days i.e., less than 12 weeks which is why no data was collected for any outcome measure.
Arm/Group | Celliant Sock | Control Sock
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Complete Wound Closure
Description: To compare the incidence of complete wound closure as defined as skin reepithelialization without drainage.
Time Frame: 12 weeks
Population: as for outcome 1
Arm/Group | Celliant Sock | Control Sock
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Number of Patients With Maintained Wound Closure
Description: The number of patients with maintained wound closure.
Time Frame: 3 months
Population: as for outcome 1
Arm/Group | Celliant Sock | Control Sock
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 79 days
Description: No subject was assigned to the Control arm and this study was terminated.
Arm/Group | Celliant Sock | Control Sock
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study records and results will be owned by the institution. Any medical records from the study will remain the property of the institution. The Institution is The University of Texas Southwestern Medical Center.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT04709419/Prot_SAP_000.pdf